CLINICAL TRIAL: NCT05963646
Title: Optical Coherence Tomography and Microperimetry Biomarker Evaluation in Patients With Geographic Atrophy Study
Acronym: OMEGA
Status: Completed | Type: Observational
Sponsor: Institute of Molecular and Clinical Ophthalmology Basel (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: OMEGA
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Age-Related Macular Degeneration; Geographic Atrophy; Visual Field Defect, Central Scotoma of Both Eyes
Keywords: Microperimetry; Fundus-controlled perimetry
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Natural history study — Patients were monitored with a panel of visual function tests and imaging modalities. Functional tests included best-corrected visual acuity (BCVA), low-luminance visual acuity (LLVA), and contrast sensitivity function evaluation (qCSF method). Imaging assessments included fundus autofluorescence, optical coherence tomography and optical coherence tomography angiography.

SUMMARY:
This study is a biomarker evaluation study in patients with geographic atrophy secondary to age-related macular degeneration (AMD). The study evaluates microperimetry (fundus-controlled perimetry) and optical coherence tomography imaging for assessing changes in retinal sensitivity and anatomy over time.

DETAILED DESCRIPTION:
The optical coherence tomography (OCT) and microperimetry biomarker evaluation in patients with GA (OMEGA) study aims to systematically compare a panel of established and novel visual function and structural outcome measures for monitoring GA progression. This prospective, natural-history study was performed at a tertiary referral center (University Hospital Basel, PI: Prof. Dr. med. Hendrik P.N. Scholl). The study included a baseline visit and follow-up visits at weeks 12, 24, and 48.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the study
2. Age >60 years
3. Ability (including a sufficient general health status according to investigators judgement) and willingness to undertake all scheduled visits and assessments including predefined methodology and standards utilizing microperimetry
4. GA secondary to AMD with no evidence of prior or active choroidal neovascularization (CNV) in the study eye
5. GA lesion in the study eye must reside completely within the FAF imaging field (Field 2-30 degree image centered on the fovea)
6. BCVA of 20/63 or better (Snellen equivalent) using ETDRS charts at starting distance of 4 m in the study eye
7. Well demarcated area(s) of GA secondary to AMD with no evidence of prior or active CNV in the study eye. The total GA lesion size >1.2 mm2 (approximately >0.5 disc area [DA]) and <17.78 mm2 (approximately <7 DA) and must reside completely within the FAF imaging field (Field 2, i.e., 30 degree image centered on the fovea). If GA is multifocal, at least 1 focal lesion must be >1.2 mm2 (approximately >0.5 DA).
8. Sufficiently clear ocular media, adequate pupillary dilation, and fixation to permit quality fundus imaging in the study eye.

Exclusion Criteria:

1. GA in either eye due to causes other than AMD (for example, monogenetic macular dystrophies [e.g., Stargardt disease, cone rod dystrophy] or toxic maculopathies [e.g., chloroquine/hydroxychloroquine maculopathy])
2. Receiving active treatment in any studies of investigational drugs for GA/dry AMD in the study eye
3. Mean sensitivity difference > 3 dB between the two microperimetry examinations in the screening visit.
4. History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye
5. Previous laser photocoagulation for CNV, diabetic macular edema, retinal vein occlusion, and proliferative diabetic retinopathy in the study eye
6. Prior treatment with Visudyne, external-beam radiation therapy, or transpupillary thermotherapy in the study eye
7. History of prophylactic subthreshold laser treatment for AMD in the study eye
8. Previous intravitreal drug delivery in the study eye (e.g., intravitreal corticosteroid injection, anti-angiogenic drugs, anti complement agents, or device implantation). A single intraoperative administration of a corticosteroid during cataract surgery for cystoid macular edema prophylaxis at least 3 months prior to screening is permitted.
9. RPE tear that involves the macula in either eye
10. Any concurrent ocular or intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could do either of the following:

    * Require medical or surgical intervention during the study period to prevent or treat vision loss that might result from that condition
    * If allowed to progress untreated, could likely contribute to loss of at least two Snellen equivalent lines of BCVA during the study period
11. Previous violation of the posterior capsule in the study eye unless it occurred as a result of Yttrium Aluminum Garnet (YAG) laser posterior capsulotomy in association with prior posterior chamber intraocular lens implantation

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with manifest geographic atrophy (total GA lesion size >1.2 mm2) secondary to age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in retinal sensitivity in the junctional zone | Week 12
  Change from baseline in retinal sensitivity in the junctional zone and in the perilesional zone of the largest atrophic loci as assessed by microperimetry
Change in retinal pigment epithelium (RPE) thickness in the junctional zone | Week 12
  Change from baseline in retinal pigment epithelium (RPE) layer thickness in the junctional zone and in the perilesional zone measured by OCT
Change in photoreceptor thickness in the junctional zone | Week 12
  Change from baseline in photoreceptor layer thickness in the junctional zone and in the perilesional zone measured by OCT

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Holz FG, Bindewald-Wittich A, Fleckenstein M, Dreyhaupt J, Scholl HP, Schmitz-Valckenberg S; FAM-Study Group. Progression of geographic atrophy and impact of fundus autofluorescence patterns in age-related macular degeneration. Am J Ophthalmol. 2007 Mar;143(3):463-72. doi: 10.1016/j.ajo.2006.11.041. Epub 2006 Dec 22. PMID 17239336
- [Background] Pfau M, Muller PL, von der Emde L, Lindner M, Moller PT, Fleckenstein M, Holz FG, Schmitz-Valckenberg S. MESOPIC AND DARK-ADAPTED TWO-COLOR FUNDUS-CONTROLLED PERIMETRY IN GEOGRAPHIC ATROPHY SECONDARY TO AGE-RELATED MACULAR DEGENERATION. Retina. 2020 Jan;40(1):169-180. doi: 10.1097/IAE.0000000000002337. PMID 30300264
- [Background] Pfau M, von der Emde L, de Sisternes L, Hallak JA, Leng T, Schmitz-Valckenberg S, Holz FG, Fleckenstein M, Rubin DL. Progression of Photoreceptor Degeneration in Geographic Atrophy Secondary to Age-related Macular Degeneration. JAMA Ophthalmol. 2020 Oct 1;138(10):1026-1034. doi: 10.1001/jamaophthalmol.2020.2914. PMID 32789526
- [Result] Ansari G, Scharer N, Camenzind Zuche H, Gabrani C, Anders P, Pfau K, Valmaggia P, Giani A, Esmaeelpour M, Chingning Yamaguchi T, Prunte CF, Maloca PM, Schmetterer L, Scholl HPN, Pfau M. The Optical Coherence Tomography and Microperimetry Biomarker Evaluation in Patients with Geographic Atrophy (OMEGA) Study: Design and Baseline Characteristics - OMEGA Report 1. Ophthalmic Res. 2023;66(1):1392-1401. doi: 10.1159/000535375. Epub 2023 Nov 28. PMID 38016431